CLINICAL TRIAL: NCT01874301
Title: Evaluation of Changes in Gut Transit Time and Gastrointestinal Symptoms Following the Consumption of a Probiotic Food Product in Adults With Constipation
Brief Title: Probiotics and Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12.05.NRC
Record Dates: First submitted 2013-05-31; First posted 2013-06-11 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High quantity probiotic food product (Experimental)
  Interventions: Other: High quantity probiotic
- Low quantity probiotic food product (Experimental)
  Interventions: Other: Low quantity probiotic
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: High quantity probiotic — The intervention type is food product
  Arms: High quantity probiotic food product
Other: Low quantity probiotic — The intervention type is food product
  Arms: Low quantity probiotic food product
Other: placebo
  Arms: Placebo

SUMMARY:
Gastrointestinal discomfort regularly affects >25% of the population worldwide. One of the major contributors to Gastrointestinal discomfort is constipation, which has a prevalence of ~15%, and symptoms of which have a significant negative impact on the sufferer's quality of life. One of the hallmarks of chronic constipation is slow progression of contents through the gut (i.e. slow gut / colonic transit time), which may be associated with hard stools that are difficult to expel. Previous studies have shown that probiotics improve colonic transit times in constipated patients. In addition, several other studies, employing a range of different probiotic strains, have shown a significant increase in defaecation frequency and improvement in stool consistency. However, the clinical relevance of these results is uncertain, due to small sample sizes and limitations in study methodology. The current study is designed to compare changes in gut transit time and gastrointestinal symptoms following 4 weeks consumption of a probiotic strain in a randomized, double-blind, placebo-controlled manner, in adults with constipation.

DETAILED DESCRIPTION:
This is an adaptive, parallel, double-blinded, randomized, placebo-controlled, stratified clinical study, comparing three study arms (two quantities of the probiotic active component and one placebo)with equal allocation ratio. Recruitment of subjects to the low quantity of the probiotic will be after fulfilling certain criteria at interim. After half of the subjects in the two study groups of high quantity and placebo have completed the study (40 subjects), an interim analysis will be performed. Depending on the observed effect size and the conditional power, the study may be stopped for futility, continued with the two groups or continued with inclusion of the third group of low dose probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women
* female subjects of child-bearing potential must be willing to use a reliable method of contraception throughout the study period
* Age 18 - 65
* BMI: 18.5 - 29.9 kg/m2
* Symptoms of constipation for a minimum of 3 months
* Recruitment based on simplified core ROME III diagnostic criteria for functional constipation (based on specific screening questions):a). average Bristol stool type of 1 - 4 AND frequency of 1 - 3 spontaneous bowel movements (SBMs) per week b). plus at least ONE of: straining on at least 25% of defaecations; sensation of incomplete evacuation on at least 25% of defaecations; sensation of anorectal obstruction / blockage on at least 25% of defaecations; use of manual manoeuvres on at least 25% of defaecations.
* Cleveland Clinic constipation score (CCCS) of 8-15
* Willing and able to consume a milk-based product daily for 4 weeks
* Low-moderate fibre intake (≤18g) determined by the semi-quantitative food intake screener known as the Block Fibre Screener
* No regular use of fibre supplementation (e.g. Fybogel, Lactulose) over the week prior to the screening visit, and no more than 6 standard doses in the past 1 month prior to the screening visit. Also, willing to discontinue fibre supplementation and other probiotics, prebiotics, fermented milk, yoghurt or laxatives at least 2 weeks prior to and during the consumption phase and the follow-up phase
* Ability to understand the patient information sheet and instructions in English, and able to provide informed consent

Exclusion Criteria:

* Subjects who report lactose intolerance and/or are allergic to cow milk protein or soya
* Regular consumption of probiotics, fibre supplements (including prebiotics), fermented milk, yogurt, laxatives, or those unwilling to discontinue these at least 2 weeks prior to and during the study
* Pregnant or breast-feeding women
* Ongoing other diagnosed gastrointestinal disease or complication (e.g. IBS, Crohn's disease, Coeliac disease, chronic diarrhoea, etc.)
* Any clinical relevant abnormalities in the screening visit medical examination or alarm features such as sudden unintentional weight loss, rectal bleeding, recent change in bowel habit (<3 months), abdominal pain and stool positive for occult blood
* Prior abdominal surgery (including gastric bypass or laparoscopic banding), except cholecystectomy and appendicectomy
* Neurologic diseases such as multiple sclerosis, stroke, spinal cord injury, Hirschsprung disease
* Ongoing therapy with drugs known to affect gut motility, such as prokinetic agents (such as metoclopramide, domperidone, erythromycin, azithromycin), anti-emetic agents, anxiolytics (such as benzodiazepines), antidepressive agents (such as trycyclics, SSRI's etc.), narcotic analgesic agents (such as methadone, fentanyl), anticholinergic agents for IBS, medications for constipation (including enemas, cathartics, polyethylene glycol solutions), 5HT3 antagonists, anti-diarrheal agents (such as loperamide), opiate agents used to treat diarrhoea, NSAIDs (more than once daily), other antibiotics taken during or within 4 weeks of study onset, magnesium-containing antacids
* Illness that may preclude the subject's ability to complete the study or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness, severe cardiovascular disease, chronic renal failure or eating disorders) or any other serious illness resulting in >2 weeks inability to work in the 3 months before the study start
* Subjects with co-morbid illnesses such as cardiovascular, endocrine, renal or other chronic disease likely to affect gut motility or limit normal functions (e.g. reduced mobility or increased fragility)
* HADS score of >11
* Ongoing alcohol, drug, or medication abuse
* Self-reported symptoms of pelvic organ prolapse
* Moderate or severe active local anorectal problems such as recurrent anal fissures, bleeding, large prolapsing haemorrhoids, etc
* Participation in another study with any investigational product within 3 months of screening
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time- 2 groups | After 2 weeks consumption of the study product
  To evaluate change in whole gut transit time 2 weeks after consumption of the study product in constipated patients consuming the study product containing probiotics in high quantity, compared to those consuming placebo

SECONDARY OUTCOMES:
Regional colonic transit time- all groups | After 2 weeks consumption of the study product
  To evaluate change in the regional (right colon, left colon, and rectosigmoid)transit time 2 weeks after consumption of the study product in all groups
Whole gut and Regional colonic transit time- all groups | After 4 weeks consumption of the study product
  To evaluate the whole gut and regional colonic transit time after 4 weeks consumption of the study product in all study groups
Whole gut transit time- all groups | After 2 weeks consumption of the study product
  To evaluate change in whole gut transit time 2 weeks after consumption of the study product in all groups
Response to the Patient assessment of constipation symptoms (PAC-SYM) - all groups | After 2&4 weeks consumption of the study product
  To evaluate change in Gastrointestinal symptoms 2&4 weeks after consumption of the study product in all groups
Cleveland Clinic constipation score - all groups | After 1&2&4 weeks consumption of the study product
  To evaluate change in Gastrointestinal symptoms 2&4 weeks after consumption of the study product in all groups
Stool frequency- all groups | After 2&4 weeks consumption of the study product
  Assessed through daily bowel diary records for each bowel movement
Stool consistency - all groups | After 2&4 weeks consumption of the study product
  To evaluate stool form (Bristol stool scale) 2&4 weeks after consumption of the study product in all groups
Response to the constipation quality of life (PAC-QOL)questionnaires - all groups | After 2&4 weeks consumption of the study product
  To evaluate change in quality of life 2&4 weeks after consumption of the study product in all groups
Tolerance to the study product- all groups | After 2&4 weeks consumption of the study product
  Response to tolerance questionnaire 2&4 weeks after consumption of the study product in all groups
Global Constipation Symptom Score - all groups | After 1&2&4 weeks consumption of the study product
  To evaluate change in Gastrointestinal symptoms 2&4 weeks after consumption of the study product in all groups
Ease of passage - all groups | After 2&4 weeks consumption of the study product
  Assessed through daily bowel diary records for each bowel movement

OTHER OUTCOMES:
Correlation between lifestyle, diet and blood/stool biomarkers with gut function and symptoms- all groups | After 2&4 weeks consumption of the study product
  To evaluate correlation between lifestyle, diet and blood/stool biomarkers with gut function and symptoms, 2&4 weeks after consumption of the study product in all groups
Long-term changes in gut function and gastrointestinal symptoms | After 4 weeks follow-up (week 8)
  To assess long-term changes in gut function and gastrointestinal symptoms 4 weeks after the end of the study product consumption period in all study groups
Adverse Events | Through the study product consumption period (4 weeks)
  Adverse events assessed as treatment emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Scott, PhD, Principal Investigator — Wingate Institute, Queen Mary University of London
Locations (1):
- Wingate Institute, Queen Mary University of London, London, United Kingdom